CLINICAL TRIAL: NCT05648591
Title: Open-label Safety Study of a 1-year 8 to 24 mg/Day Dose Regimen of Iloperidone (FANAPT®) in Adolescent Patients With Schizophrenia or Bipolar I Disorder
Brief Title: Safety and Tolerability of Open-Labeled Iloperidone in Adolescents
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VYV-683-4101
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: fanapt
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iloperidone (Experimental): Open-label iloperidone
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone — oral tablet
  Other Names: VYV-683; FANAPT

SUMMARY:
To evaluate the safety and tolerability of iloperidone in adolescent patients with schizophrenia or bipolar I disorder for up to 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide assent and willing to complete all aspects of the study
* Patient's parent or legal guardian willing and able to provide consent
* Male or female patients 12 through 17 years of age (inclusive)
* Clinical diagnosis of either schizophrenia or bipolar I disorder

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* A positive test for drugs of abuse

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) in the treatment period. | 1 year

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Decatur, Georgia
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Garfield Heights, Ohio
  - Vanda Investigational Site, Westlake, Ohio
  - Vanda Investigational Site, Everett, Washington